CLINICAL TRIAL: NCT05780645
Title: A Two-Part Phase 1 Study to Evaluate the Pharmacokinetic Profile of ALXN2050 Modified Release Prototype Formulations and Immediate Release Reference Tablet in Healthy Adult Participants
Brief Title: A Study to Investigate the Pharmacokinetic Profile of ALXN2050 Modified Release Prototype Formulations and Immediate Release Reference Tablet in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7841C00008
Record Dates: First submitted 2023-03-13; First posted 2023-03-22 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Healthy Participants
Keywords: Healthy participants
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Regimen A: Participants will receive Dose B (3 x Dose A) ALXN2050 IR Tablet orally under fasted conditions.
  Regimen B: Participants will receive Dose C ALXN2050 MR Prototype Tablet orally under fasted conditions.
  Optional Regimens C, D, E, and F
  Interventions: Drug: ALXN2050 MR Prototype Tablet; Drug: ALXN2050 Immediate Release (IR) Tablet
- Cohort 2 (Experimental): Regimen G: Participants will receive Dose B (3 x Dose A) ALXN2050 IR Tablet orally under fasted conditions.
  Regimen H: Participants will receive Dose C ALXN2050 MR Prototype Mini-Tablet orally under fasted conditions.
  Optional Regimens: I, J, K, and L
  Interventions: Drug: ALXN2050 Immediate Release (IR) Tablet; Drug: ALXN2050 MR Prototype Mini-Tablet

INTERVENTIONS:
Drug: ALXN2050 MR Prototype Tablet — Participants will receive various doses of the MR Prototype Tablet orally.
  Arms: Cohort 1
Drug: ALXN2050 Immediate Release (IR) Tablet — Participants will receive a single dose IR (ALXN2050 Film Coated Tablet) tablet orally.
Drug: ALXN2050 MR Prototype Mini-Tablet — Participants will receive various doses of the MR Prototype Mini-Tablet orally.
  Arms: Cohort 2

SUMMARY:
The primary objectives of this study are to investigate the relative bioavailability and PK (Pharmacokinetic) profile of 2 ALXN2050 MR (Modified Release) formulations in comparison with the IR (Immediate Release) formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating healthy females.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical or neurological examination, vital signs, 12-lead ECG, screening clinical laboratory profiles (hematology, biochemistry, coagulation, and urinalysis), as deemed by the Investigator or designee.
* BMI within the range of 18.0 to 30.0 kg/m2 (inclusive), with a minimum body weight of 50.0 kg at screening.
* Female participants of childbearing potential and male participants must follow protocol-specified contraception guidance.

Exclusion Criteria:

* History of clinically significant respiratory, cardiovascular, dermatological, hepatic, renal, GI, endocrinological, hematological, psychological, psychiatric, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* History of meningococcal infection.
* History of clinically significant hypersensitivity reactions to commonly used antibacterial agents, including beta lactams, penicillin, aminopenicillins, fluoroquinolones (specifically including ciprofloxacin), cephalosporins, and carbapenems, which in the opinion of the Investigator would make it difficult to properly provide either empiric antibiotic therapy or treat an active infection.
* History of clinically significant hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
* History of significant multiple and/or severe allergies (eg, drug, latex allergy, band aids, adhesive dressing, or medical tape). Hay fever is allowed unless it is active.
* History of seizures including childhood seizures.
* History of significant head injury, or head trauma requiring medical evaluation.
* History of malignancy within 5 years of screening, with the exception of non-melanoma skin cancer or carcinoma in situ of the cervix that has been treated with no evidence of recurrence.
* Any previous procedure, including history of stomach or intestinal surgery or resection, cholecystectomy, gallstones, TIPS, or surgical shunt, that could alter absorption or excretion of orally administered drugs.
* Significant current or chronic history of liver disease.
* Known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ALXN2050 | Up to 96 hours postdose
Time to Reach Cmax (Tmax) of ALXN2050 | Up to 96 hours postdose
Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of Last Measurable Concentration (AUC0-last) of ALXN2050 | Up to 96 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Day 1 up to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Ruddington, United Kingdom